CLINICAL TRIAL: NCT03463694
Title: Edinburgh and Lothian Virus Intervention Study in Kids (ELVIS Kids): A Randomised Controlled Trial of Hypertonic Saline Nose Drops in Children With Upper Respiratory Tract Infections
Brief Title: Edinburgh and Lothian Virus Intervention Study in Kids
Acronym: ELVIS Kids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ELVIS Kids
Record Dates: First submitted 2018-02-14; First posted 2018-03-13 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Upper Respiratory Tract Infections; Virus; Virus Shedding; Pediatric ALL
MeSH Terms: conditions — Respiratory Tract Infections; Virus Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: ELVIS Kids is a parallel, open label, randomised controlled trial (RCT) of HS nose drops (~2.6% NaCl) vs. standard care in children <7 years of age with symptoms of an URTI.
Who Masked: Outcomes Assessor
Masking Description: The team in the virology lab carrying out the analysis of the nasal swabs will be blinded to the allocation of the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertonic Saline ~2.6% NaCl (Experimental): 3 drops each nostril of Hypertonic Saline (HS) at least 4 times a day until asymptomatic or maximum of 28 days
  Interventions: Other: Na Cl solution
- Standard Care (No Intervention): Control arm of standard symptomatic care only

INTERVENTIONS:
Other: Na Cl solution — ~2.6% NaCl solution prepared from sea salt
  Arms: Hypertonic Saline ~2.6% NaCl

SUMMARY:
ELVIS Kids is a parallel, open label, randomised controlled trial (RCT) of Hypertonic Saline (HS) nose drops (~2.6% NaCl) vs. standard care in children <7 years of age with symptoms of an Upper Respiratory Tract Infection (URTI).

DETAILED DESCRIPTION:
The study will run over ~30 months. Children are recruited prior to, or within 48 hours of developing URTI symptoms by advertising in areas such as local schools, nurseries, health centres and workplaces as well as social media. For the purposes of this study an URTI is defined as: at least two respiratory symptoms (nasal stuffiness, runny nose, cough, sore throat, or sneezing) OR one respiratory symptoms and at least one systemic symptom (lethargy, muscle pain, headache, pyrexia ≥38°C).

Willing parents/guardians, of children <7 years of age, will be directed by the study advertising to contact the research team at their local research site if they are interested in participating. Children will be randomised to either a Control arm of standard symptomatic care, or an Intervention arm of 3 drops each nostril of HS at least 4 times a day until 24 hours after asymptomatic or maximum of 28 days. All participants will be requested to obtain a mid-turbinate nasal swab prior to first nasal HS drops (repeated daily for 5 days), a daily symptom diary (CARIFS, a valid illness measure in the UK), and an end of illness questionnaire (healthcare use, adverse events, acceptability, infection in household contacts, parental time taken off usual activities). Parent/guardian of the children allocated to the intervention arm will be taught how to prepare the HS. Parent/guardian of children who are asymptomatic at recruitment are requested to inform CCRF when the child develops an URTI (within 48 hours) and follow the instructions already provided to them when given the go-ahead to start the trial. On day 28, parents/guardians will be contacted to determine if their child suffered from wheeze either during the illness or at any point until day 28. Participation in the study will end on day 28.

ELIGIBILITY:
INCLUSION CRITERIA

1. Children between corrected gestational age of ≥40 weeks and <7 years of age
2. Children without URTI OR ≤48 hours of URTI* starting.

   * A URTI being defined as at least two respiratory symptoms (nasal congestion (i.e. stuffy nose), runny nose, cough, sore throat) OR one respiratory symptom + at least one systemic symptom (Low energy/tired, muscle aches/pains, headache, fever ≥38°C).

EXCLUSION CRITERIA

1. Children needing immediate medical attention
2. Children using saline drops/sprays at the time of randomisation
3. Children on immunosuppressive medication, regular oral/inhaled steroids, regular antibiotics (use of antibiotics is allowed as long as the child does not need regular antibiotics)
4. Children with a known chronic illness (e.g. cystic fibrosis, cardiac, renal, liver, lung, neurological conditions) apart from wheeze or asthma which are not exclusions if the child is otherwise well and not on regular steroids)
5. Children being followed up for developmental delay
6. Children receiving the nasal flu vaccine ≤14 days ago
7. Children taking part in another interventional trial
8. If parents/guardians indicating that they are unable to comply with the study protocol prior to randomisation
9. If parents/guardians are unable to understand written or spoken English
10. Children randomised to ELVIS KIDS on a previous episode of URTI
11. Children with a concurrently participating sibling

Ages: 40 Weeks to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 407 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Time to the first report that the child is "not unwell". | Maximum of 28days
  Time until child not unwell

SECONDARY OUTCOMES:
Severity of all symptoms | 1-28 days (or until child is well)
  Recorded by parents from options: No Problem, Minor Problem,Moderate Problem,Major Problem or Unknown/Not Applicable
The length of time for individual symptoms to resolve | 1-28 days (or until child is well)
  Recorded as: No Problem, Minor Problem,Moderate Problem,Major Problem or Unknown/Not Applicable
Severity of individual symptoms | 1-28 days (or until child is well)
  Recorded by parents from options: No Problem, Minor Problem,Moderate Problem,Major Problem or Unknown/Not Applicable
Contacting healthcare (NHS 24, OOH, GP) -Number of participants | 1-28 days (or until child is well)
  Number of participants
Contacting healthcare (NHS 24, OOH, GP) -Frequency of contacts | 1-28 days (or until child is well)
  Number of contacts
Participants needing GP appointments- Number of participants | 1-28 days (or until child is well)
  Number of appointments
Participants needing GP appointments- Frequency of contacts | 1-28 days (or until child is well)
  Number of appointments
Number of participants attending hospital and diagnosis - Number of participants | 1-28 days (or until child is well)
  Number of participants
Number of participants attending hospital and diagnosis - Frequency of contacts | 1-28 days (or until child is well)
  Number of attendances
Length of stay in hospital if admitted | 1-28 days (or until child is well)
  Length in Days
Number of participants reporting wheeze during illness and between end of illness to 28 days | Day 28
  Number reporting wheeze
Number of participants reporting over the counter medication use | 1-28 days (or until child is well)
  Number of participants
Duration of viral shedding | Days 1-5
  Viral shedding duration in days
Reduction in viral shedding | Days 1-5
  Log conversion of each positive result will be done using the following formula: (40-CT of specimen)/3.3 to estimate change in shedding.
Rate of reduction in viral shedding | Days 1-5
  Rate of viral shedding duration in days
Reduction in transmission to household contacts | 1-28 days (or until child is well)
  Questionnaire - reported number of adults and children catching URTI
Number of participants reporting side effects of nasal drops | 1-28 days (or until child is well)
  Side effects reported
Types and severity of side effects reported | 1-28 days (or until child is well)
  Side effects reported
Number of days lost from school/nursery for child | 1-28 days (or until child is well)
  Number of days
Number of days lost from work for parent/guardian | 1-28 days (or until child is well)
  Number of days
Cost of over the counter medication used | 1-28 days (or until child is well)
  Cost of medicine used.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Ramalingham, Principal Investigator — NHS Lothian
Locations (1):
- Childrens' Clinical Research Facility, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ramalingam S, Graham C, Oatey K, Rayson P, Stoddart A, Sheikh A, Cunningham S; ELVIS Kids Trial Investigators. Study protocol of the Edinburgh and Lothian Virus Intervention Study in Kids: a randomised controlled trial of hypertonic saline nose drops in children with upper respiratory tract infections (ELVIS Kids). BMJ Open. 2021 May 5;11(5):e049964. doi: 10.1136/bmjopen-2021-049964. PMID 33952557